CLINICAL TRIAL: NCT00246038
Title: A Phase II Evaluation of the Safety and Efficacy of the Boston Scientific ENOVUS AAA Endograft in the Treatment of Abdominal Aortic Aneurysms
Brief Title: The Boston Scientific ENOVUS Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor cancelled the development program, and never conducted the study.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Pamela Grady, PhD, Director, Clinical Programs, Boston Scientific Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810-0001
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; Aortic Aneurysm; AAA; Endovascular; Stent Graft; Endograft; Vascular Prostheses
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Boston Scientific ENOVUS AAA Endograft

SUMMARY:
A prospective, actively controlled, consecutively enrolling, non-randomized multi center clinical evaluation of the safety and efficacy of the Boston Scientific ENOVUS AAA Endograft when used in the treatment of patients with AAA (Treatment Group) as compared to patients treated with conventional open surgery (Control Group).

DETAILED DESCRIPTION:
The primary objectives of this study are to determine whether the Boston Scientific ENOVUS AAA Endograft is a safe and effective method of treating AAA's in those patients considered to be suitable candidates for open surgical repair. The safety of the Boston Scientific ENOVUS AAA Endograft will be determined by comparing the rate of major morbidity in the Treatment Group against the rate of major morbidity in the Control Group within 30 days of the initial procedure. The efficacy of the Boston Scientific ENOVUS AAA Endograft will be determined by evaluating the proportion of patients in the Treatment Group that are free from AAA rupture and conversion to open surgical repair within 1 year of the initial procedure.

The secondary safety endpoints will be compared between the Treatment and Control Groups:Mortality rates at 30 days and 1 year, AAA related mortality at 30 days and 1 year. The secondary efficacy endpoints will be evaluated in the Treatment Group only and include: Technical success, enlargement of AAA, migration, significant endoleak, and loss of device integrity. Secondary Clinical Utility endpoints will be compared between the Treatment and Control groups and will include: blood loss, duration of procedure, ICU stay, length of hospital stay, and duration of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet all of the following inclusion criteria to be eligible for enrollment into this study:

  1. Patient is > 18 years of age
  2. Females of childbearing potential have a negative pregnancy test at the time of treatment
  3. Patient has signed an Institutional Review Board (IRB) approved Informed Consent Form
  4. Patient is considered by the treating physician to be a candidate (i.e., categories I, II, or III) for elective open surgical repair of the AAA per American Society of Anesthesiology (ASA) refer to Appendix II. ASA grade IV patients may be enrolled provided their life expectancy is greater than 1 year.
  5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:•Abdominal aortic aneurysm >4.5 cm in diameter

     * Aneurysm has increased in size by 0.5 cm in last 6 months.
     * Maximum diameter of aneurysm exceeds one and one-half times the transverse dimension of an adjacent normal aortic segment
  6. Patient must be willing to comply with all required follow-up exams (open surgical control patients are followed through one year, Treatment Group patients are followed through five years in the study with lifelong follow up by physician thereafter).

Exclusion Criteria:

* Patients that meet ANY of the following are not eligible for enrollment into the study:

  1. Aneurysm dissection
  2. Acutely ruptured aneurysm
  3. Acute vascular injury
  4. Need for emergent surgery
  5. Patient has a known thoracic aortic aneurysm or dissection.
  6. Patient has unstable angina (defined as angina characterized by progressive increase in anginal symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
  7. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
  8. Patient has history of bleeding disorders or refuses blood transfusions.
  9. Patient has baseline serum creatinine level >2.0 mg/dl
  10. Patient has a known hypersensitivity or contraindication to anticoagulation that is not amenable to pre-treatment.
  11. Patient has a mycotic aneurysm or has an active systemic infection
  12. Patient is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta
  13. Patient has a limited life expectancy of less than 1 year
  14. Patient is currently participating in another investigational device or drug clinical trial
  15. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving this treatment, pre-treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Efficacy will evaluate patients (Treatment Group) free from AAA rupture and surgical conversion within 1 year of the initial procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A. White, MD; Chief, Vascular Surgery, Principal Investigator — University of California, Los Angeles; W. Anthony Lee, MD; Assistant Professor of Surgery, Principal Investigator — University of Florida